CLINICAL TRIAL: NCT04781647
Title: A Randomized Phase 2a, Multicenter, Open-label Study Evaluating ABI-H0731-Containing Regimens in Patients With Chronic Hepatitis B
Brief Title: A Study Evaluating ABI-H0731-containing Regimens in Chinese Participants With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ABI-H0731-203 was terminated early by the study Sponsor for strategic reasons to prioritize research and development efforts on finite and curative HBV therapies.
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-H0731-203
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Chronic Hepatitis B
Keywords: cHBV; HBV; vebicorvir; VBR
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ABI-H0731 + ETV (Active Comparator): Participants with cHBV will receive ABI-H0731 with ETV for 48 weeks, followed by ETV alone for 12 weeks
  Interventions: Drug: ABI-H0731; Drug: ETV
- ABI-H0731 + ETV + Peg-IFNα (Experimental): Participants with cHBV will receive ABI-H0731 with ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks
  Interventions: Drug: ABI-H0731; Drug: ETV; Biological: Peg-IFNα
- ETV + Peg-IFNα (Active Comparator): Participants with cHBV will receive ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks
  Interventions: Drug: ETV; Biological: Peg-IFNα

INTERVENTIONS:
Drug: ABI-H0731 — Participants will receive ABI-H0731 300 mg tablets orally once daily
  Other Names: Vebicorvir
  Arms: ABI-H0731 + ETV; ABI-H0731 + ETV + Peg-IFNα
Drug: ETV — Participants will receive ETV 0.5 mg tablets orally once daily
  Other Names: Entecavir
Biological: Peg-IFNα — Participants will receive Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
  Other Names: Pegylated-interferon Alpha
  Arms: ABI-H0731 + ETV + Peg-IFNα; ETV + Peg-IFNα

SUMMARY:
The purpose of this study is to evaluate the safety, antiviral activity, and pharmacokinetics of ABI-H0731 in combination with entecavir (ETV) and with ETV plus pegylated-interferon alpha (Peg-IFNα) in Chinese participants with chronic hepatitis B virus infection (cHBV)

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 36 kg/m^2 and a minimum body weight of 45 kg (inclusive)
* Female subjects must be non-pregnant and have a negative serum pregnancy test
* Chronic hepatitis B infection, defined as HBV infection for ≥6 months documented, for example, by at least 2 measurements of HBsAg positivity and/or detectable HBV DNA ≥6 months apart (inclusive of Screening). For subjects without clear documentation of CHB, serum immunoglobulin M (IgM) antibody to the HBV core antigen (HBcAb) must be negative at Screening to exclude acute HBV infection.
* HBeAg positive with HBV DNA ≥2 × 10^4 IU/mL at Screening
* Lack of cirrhosis or advanced liver disease
* A candidate for interferon-based therapy
* Agreement to comply with protocol-specified contraceptive requirements
* Agreement to abstain from alcohol abuse and the use of illicit substances from Screening through the duration of the study
* In good general health, except for cHBV, in the opinion of the Investigator
* Able to take oral medication and be willing to receive subcutaneous injections of Peg-IFNα.

Exclusion Criteria:

* Current or prior treatment for CHB with

  * A nucleos(t)ide reverse transcriptase inhibitor of the HBV polymerase (NrtI) (ETV, tenofovir disoproxil fumarate or tenofovir alafenamide) for >4 weeks at any time. Note, NrtI treatment of ≤4 weeks duration cannot be within 6 months prior to Screening
  * Interferon-based therapy within 6 months prior to Screening
  * Liver-protecting and/or ALT-lowering treatment including traditional Chinese medicine within 1 month of Screening
  * Lamivudine, telbivudine or adefovir (of any duration)
  * Previous treatment with siRNA within 9 months prior to Screening
  * HBV core inhibitors (any duration)
  * Previous treatment with any other investigational agent for HBV infection within 6 months prior to Screening
* Co-infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV) hepatitis C virus (HCV), hepatitis E virus (HEV), or hepatitis D virus (HDV)
* Females who are lactating, or wish to become pregnant during the course of the study
* History or evidence of advanced liver disease or hepatic decompensation at any time prior to, or at the time of Screening
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to Screening
* Clinically significant psychiatric disease, including severe depression, history of suicidal ideation or suicide attempt
* Clinically significant cardiac disease including poorly controlled or unstable hypertension; pulmonary disease; chronic or recurrent renal or urinary tract disease; liver disease other than cHBV; endocrine disorder; autoimmune disorder; poorly controlled diabetes mellitus; neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment; seizure disorders requiring treatment; ongoing infection or other medical conditions requiring frequent medical management; or pharmacologic or surgical treatment that, in the opinion of the Investigator or the Sponsor, makes the subject unsuitable for study participation
* History of hepatocellular carcinoma (HCC)
* History of malignancy other than HCC unless the subject's malignancy has been in complete remission off chemotherapy and without additional medical or surgical interventions during the 3 years before Screening
* History or presence at Screening of electrocardiogram (ECG) abnormalities deemed clinically significant, in the opinion of the Investigator
* History of hypersensitivity or idiosyncratic reaction to any components or excipients of the investigational drug
* History of any significant food or drug-related allergic reactions such as, anaphylaxis or Stevens-Johnson syndrome
* Exclusionary laboratory results at Screening:

  * Hemoglobin <12g/dL for males or <11g/dL for females
  * Platelet count <100,000/mm^3
  * White blood cell count <2,500/mm^3
  * Absolute neutrophil count <1,500/mm^3
  * Albumin <lower limit of normal
  * History of thyroid disease poorly controlled on prescribed medications, with thyroid-stimulating hormone (TSH), free triiodothyronine or free thyroxine (T4) outside the normal limits
  * Total bilirubin >1.2 × upper limit of normal (ULN)
  * Direct bilirubin >1.2 × ULN
  * ALT ≤1 x ULN or ≥10 × ULN
  * Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at Screening is >ULN but <100 ng/mL, the participant is eligible if a hepatic imaging trial prior to initiation of study drug reveals no lesions indicative of possible HCC.
  * International Normalized Ratio >1.5 × ULN unless on a stable anticoagulant regimen
  * Glomerular filtration rate <60 mL/min/1.73 m^2 by Chronic Kidney Disease Epidemiology Collaboration equation
  * Serum creatinine >1.5 x ULN
  * Any other laboratory abnormality deemed clinically significant by the Sponsor or the Investigator.
* Subjects receiving prohibited concomitant medications or medications that should be avoided within 7 days or 5 half-lives (if known), whichever is longer, prior to administration of the first dose of study drug (Day 1) and for the duration of the study period. Please refer to Exclusion Criterion #1 for criteria regarding liver protecting and/or ALT lowering agents
* Participation in another clinical study of any non-HBV-related drug or device whereby the last investigational drug/device administration is within 60 days or 5 half-lives prior to the first study drug administration (Day 1), whichever is longer.
* Subjects who have received, in the previous 4 weeks, a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, or high-dose steroids, or other immunosuppressants).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wang, MD, Study Director — Assembly Biosciences
Locations (9):
- China (9):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanfang Hospital, First Military Medical University, Guangzhou, Guangdong
  - 8th Affiliated Hospital of Guangzhou, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin University First Hospital, Changchun, Jilin
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The first affiliated Hospital, College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ABI-H0731 + Entecavir (ETV): Participants with cHBV received ABI-H0731 with ETV for 48 weeks, followed by ETV alone for 12 weeks or until the study was early terminated
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
- ABI-H0731 + ETV + Pegylated-interferon Alpha (Peg-IFNα): Participants with cHBV received ABI-H0731 with ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks or until the study was early terminated
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
  Peg-IFNα: Participants received Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
- ETV + Peg-IFNα: Participants with cHBV received ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks or until the study was early terminated
  ETV: Participants received ETV 0.5 mg tablets orally once daily
  Peg-IFNα: Participants received Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
Period: Overall Study
Arm/Group | ABI-H0731 + Entecavir (ETV) | ABI-H0731 + ETV + Pegylated-interferon Alpha (Peg-IFNα) | ETV + Peg-IFNα
Started | 20 | 17 | 17
Completed | 6 | 5 | 6
Not Completed | 14 | 12 | 11
Not completed — Study terminated by Sponsor | 11 | 9 | 9
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Virology rebounded | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABI-H0731 + ETV: Participants with cHBV received ABI-H0731 with ETV for 48 weeks, followed by ETV alone for 12 weeks or until the study was early terminated
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
- ABI-H0731 + ETV + Peg-IFNα: Participants with cHBV received ABI-H0731 with ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks or until the study was early terminated
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
  Peg-IFNα: Participants received Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
- Total: Total of all reporting groups
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα | Total
Number analyzed (Participants) | 20 | 17 | 17 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 17 | 54
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.6) | 31 (5.8) | 34 (7.8) | 32 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 10 | 39
  Male | 5 | 3 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 17 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 17 | 17 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 20 | 17 | 17 | 54
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.51 (2.683) | 22.90 (2.407) | 23.44 (3.457) | 22.93 (2.843)
Years positive for HBV [Mean (Standard Deviation); unit: years] — Population: Some participants had an unknown number of years positive for HBV so they were not included in the analysis.
  years
    number analyzed (Participants) | 19 | 15 | 14 | 48
    (all) | 11.3 (9.23) | 11.2 (9.43) | 11.2 (8.91) | 11.3 (9.00)
HBV Genotype [Count of Participants; unit: Participants]
  Genotype A | 0 | 0 | 0 | 0
  Genotype B | 9 | 8 | 8 | 25
  Genotype C | 11 | 9 | 9 | 29
  Genotype D | 0 | 0 | 0 | 0
  Other Genotype | 0 | 0 | 0 | 0
HBV DNA (Log10 IU/mL) [Mean (Standard Deviation); unit: Log 10 IU/mL] | 8.2 (1.02) | 7.7 (1.11) | 8.1 (0.63) | 8.0 (0.96)
HBV pgRNA (Log10 U/mL) [Mean (Standard Deviation); unit: Log10 U/mL] | 6.5 (1.33) | 5.8 (1.43) | 6.5 (1.05) | 6.3 (1.30)
HBcrAg (Log10 kU/mL) [Mean (Standard Deviation); unit: Log10 kU/mL] | 5.5 (.59) | 5.0 (.71) | 5.4 (.46) | 5.3 (.62)
HBeAg (Log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 2.7 (.81) | 2.4 (.89) | 2.7 (.64) | 2.6 (.79)
HBsAg (Log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 4.5 (.39) | 4.1 (.76) | 4.3 (.53) | 4.3 (.58)
ALT (U/L) [Mean (Standard Deviation); unit: U/L] | 149 (65.0) | 138 (121.2) | 123 (58.5) | 137 (84.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Time Frame: Up to 60 weeks
Measure: Count of Participants; unit: Participants
Groups:
- ABI-H0731 + ETV: Participants with cHBV received ABI-H0731 with ETV for 48 weeks, followed by ETV alone for 12 weeks or until the study was early terminated.
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
- ABI-H0731 + ETV + Peg-IFNα: Participants with cHBV received ABI-H0731 with ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks or until the study was early terminated.
  ABI-H0731: Participants received ABI-H0731 300 mg tablets orally once daily
  ETV: Participants received ETV 0.5 mg tablets orally once daily
  Peg-IFNα: Participants received Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
- ETV + Peg-IFNα: Participants with cHBV received ETV and Peg-IFNα for 24 weeks, followed by ABI-H0731 with ETV for 24 weeks, followed by ETV alone for 12 weeks or until the study was early terminated.
  ETV: Participants received ETV 0.5 mg tablets orally once daily
  Peg-IFNα: Participants received Peg-IFNα with a starting dose of 180 µg solution by subcutaneous injection once weekly
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
Participants | 14 | 17 | 17

2. Primary Outcome: Number of Participants With Premature Discontinuation of Treatment
Time Frame: Up to 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
Participants | 18 | 17 | 11

3. Primary Outcome: Number of Participants With a Laboratory Abnormality
Time Frame: Up to 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
Participants | 19 | 16 | 17

4. Secondary Outcome: Mean Change From Baseline in HBV pgRNA
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, not all subjects reached Week 48.
Measure: Mean (Standard Deviation); unit: log10 U/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
log10 U/mL
  Week 1 | -1.3 (.51) | -1.5 (.69) | -.5 (.43)
  Week 2: number analyzed (Participants) | 20 | 16 | 17
  Week 2 | -1.6 (.58) | -1.9 (.79) | -.6 (.61)
  Week 4: number analyzed (Participants) | 19 | 16 | 17
  Week 4 | -2.0 (.72) | -2.2 (.74) | -.9 (.70)
  Week 6: number analyzed (Participants) | 19 | 16 | 17
  Week 6 | -2.3 (.87) | -2.6 (.67) | -1.6 (1.45)
  Week 8: number analyzed (Participants) | 19 | 16 | 17
  Week 8 | -2.5 (1.12) | -2.7 (.95) | -2.0 (1.75)
  Week 12: number analyzed (Participants) | 19 | 12 | 16
  Week 12 | -2.7 (1.15) | -3.0 (1.17) | -2.4 (1.72)
  Week 16: number analyzed (Participants) | 16 | 11 | 16
  Week 16 | -2.8 (1.28) | -2.9 (1.34) | -2.7 (1.68)
  Week 20: number analyzed (Participants) | 16 | 15 | 15
  Week 20 | -2.8 (1.38) | -3.0 (1.35) | -2.5 (1.61)
  Week 24: number analyzed (Participants) | 16 | 14 | 15
  Week 24 | -2.7 (1.55) | -3.3 (1.41) | -2.7 (1.67)
  Week 28: number analyzed (Participants) | 15 | 14 | 14
  Week 28 | -2.9 (1.66) | -3.0 (1.3) | -3.8 (1.63)
  Week 32: number analyzed (Participants) | 12 | 11 | 12
  Week 32 | -3.1 (1.52) | -3.0 (.99) | -3.2 (1.65)
  Week 36: number analyzed (Participants) | 8 | 8 | 10
  Week 36 | -3.3 (1.92) | -2.9 (1.04) | -3.8 (1.71)
  Week 40: number analyzed (Participants) | 9 | 7 | 10
  Week 40 | -3.1 (2.05) | -2.5 (1.13) | -3.3 (1.63)
  Week 44: number analyzed (Participants) | 7 | 5 | 7
  Week 44 | -4.0 (1.45) | -3.3 (.81) | -3.0 (2.39)
  Week 48: number analyzed (Participants) | 6 | 6 | 7
  Week 48 | -4.2 (1.13) | -2.4 (1.63) | -2.9 (1.81)

5. Secondary Outcome: Mean Change From Baseline HBV DNA
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, not all subjects reached Week 48.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
log10 IU/mL
  Week 1 | -2.1 (.64) | -2.1 (.53) | -2.2 (.51)
  Week 2: number analyzed (Participants) | 20 | 16 | 17
  Week 2 | -2.5 (.76) | -2.6 (.81) | -2.7 (.61)
  Week 4: number analyzed (Participants) | 19 | 16 | 17
  Week 4 | -3.2 (.92) | -2.9 (.70) | -3.4 (.72)
  Week 6: number analyzed (Participants) | 19 | 16 | 17
  Week 6 | -3.6 (1.07) | -3.6 (.99) | -4.0 (.94)
  Week 8: number analyzed (Participants) | 19 | 16 | 17
  Week 8 | -4.2 (1.21) | -4.1 (1.13) | -4.5 (.97)
  Week 12: number analyzed (Participants) | 19 | 12 | 16
  Week 12 | -4.9 (1.18) | -4.4 (1.00) | -5.1 (.89)
  Week 16: number analyzed (Participants) | 16 | 11 | 16
  Week 16 | -5.5 (1.06) | -5.2 (1.13) | -5.6 (.74)
  Week 20: number analyzed (Participants) | 16 | 15 | 15
  Week 20 | -5.8 (.99) | -5.6 (1.05) | -6.1 (.75)
  Week 24: number analyzed (Participants) | 16 | 14 | 15
  Week 24 | -6.0 (.94) | -6.0 (.92) | -6.5 (.67)
  Week 28: number analyzed (Participants) | 15 | 14 | 14
  Week 28 | -6.2 (.82) | -6.3 (.87) | -6.7 (.67)
  Week 32: number analyzed (Participants) | 12 | 11 | 12
  Week 32 | -6.2 (.93) | -6.2 (.94) | -6.7 (.52)
  Week 36: number analyzed (Participants) | 8 | 8 | 10
  Week 36 | -6.2 (1.05) | -6.2 (1.15) | -6.9 (.5)
  Week 40: number analyzed (Participants) | 9 | 7 | 10
  Week 40 | -6.2 (1.17) | -6.0 (1.10) | -6.7 (.63)
  Week 44: number analyzed (Participants) | 7 | 5 | 7
  Week 44 | -6.5 (1.15) | -5.8 (1.4) | -6.6 (.68)
  Week 48: number analyzed (Participants) | 6 | 6 | 7
  Week 48 | -6.7 (1.27) | -5.9 (1.16) | -6.8 (.75)

6. Secondary Outcome: Mean Change From Baseline in HBeAg
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, not all subjects reached Week 48.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
log10 IU/mL
  Week 8: number analyzed (Participants) | 19 | 16 | 17
  Week 8 | -.6 (.59) | -.8 (.61) | -.9 (.77)
  Week 12: number analyzed (Participants) | 19 | 12 | 16
  Week 12 | -.8 (.66) | -.8 (.46) | -1.1 (.74)
  Week 16: number analyzed (Participants) | 16 | 11 | 16
  Week 16 | -1.0 (.78) | -.9 (.50) | -1.2 (.73)
  Week 20: number analyzed (Participants) | 16 | 15 | 15
  Week 20 | -1.1 (.83) | -1.1 (.68) | -1.3 (.76)
  Week 24: number analyzed (Participants) | 16 | 14 | 15
  Week 24 | -1.1 (.91) | -1.2 (.73) | -1.3 (.78)
  Week 28: number analyzed (Participants) | 15 | 14 | 14
  Week 28 | -1.2 (.93) | -1.2 (.71) | -1.4 (.79)
  Week 32: number analyzed (Participants) | 12 | 11 | 12
  Week 32 | -1.4 (.87) | -1.2 (.70) | -1.5 (.83)
  Week 36: number analyzed (Participants) | 8 | 8 | 10
  Week 36 | -1.5 (.97) | -1.1 (.61) | -1.7 (.84)
  Week 40: number analyzed (Participants) | 9 | 7 | 10
  Week 40 | -1.5 (.95) | -1.2 (.65) | -1.8 (1.00)
  Week 44: number analyzed (Participants) | 7 | 5 | 7
  Week 44 | -1.8 (.83) | -1.1 (.57) | -1.9 (1.07)
  Week 48: number analyzed (Participants) | 6 | 6 | 7
  Week 48 | -1.9 (.88) | -1.1 (.55) | -2.1 (.96)

7. Secondary Outcome: Mean Change From Baseline in HBcrAg
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, not all subjects reached Week 48.
Measure: Mean (Standard Deviation); unit: log10 kU/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
log10 kU/mL
  Week 4: number analyzed (Participants) | 19 | 17 | 17
  Week 4 | -.4 (.49) | -.4 (.43) | -.3 (.36)
  Week 8: number analyzed (Participants) | 19 | 16 | 17
  Week 8 | -.6 (.59) | -.8 (.57) | -.8 (.8)
  Week 12: number analyzed (Participants) | 19 | 12 | 16
  Week 12 | -.9 (.68) | -.9 (.48) | -1.1 (.85)
  Week 16: number analyzed (Participants) | 16 | 11 | 16
  Week 16 | -1.0 (.68) | -1.0 (.57) | -1.2 (.82)
  Week 20: number analyzed (Participants) | 16 | 15 | 15
  Week 20 | -1.1 (.76) | -1.2 (.66) | -1.3 (.86)
  Week 24: number analyzed (Participants) | 16 | 14 | 15
  Week 24 | -1.2 (.81) | -1.3 (.73) | -1.4 (.88)
  Week 28: number analyzed (Participants) | 15 | 14 | 14
  Week 28 | -1.2 (.86) | -1.3 (.75) | -1.5 (.84)
  Week 32: number analyzed (Participants) | 12 | 11 | 12
  Week 32 | -1.3 (.87) | -1.2 (.65) | -1.7 (.83)
  Week 36: number analyzed (Participants) | 8 | 8 | 10
  Week 36 | -1.5 (.85) | -1.2 (.55) | -1.9 (.83)
  Week 40: number analyzed (Participants) | 9 | 7 | 10
  Week 40 | -1.6 (.97) | -1.3 (.6) | -1.9 (.93)
  Week 44: number analyzed (Participants) | 7 | 5 | 7
  Week 44 | -2.0 (.83) | -1.3 (.55) | -2.0 (1.04)
  Week 48: number analyzed (Participants) | 6 | 6 | 7
  Week 48 | -2.0 (.93) | -1.2 (.59) | -2.0 (1.01)

8. Secondary Outcome: Mean Change From Baseline in HBsAg
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, not all subjects reached Week 48.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 17
log10 IU/mL
  Week 4: number analyzed (Participants) | 19 | 17 | 17
  Week 4 | -.2 (.48) | -.1 (.39) | -.2 (.25)
  Week 8: number analyzed (Participants) | 19 | 16 | 17
  Week 8 | -.4 (.51) | -.4 (.66) | -.5 (.64)
  Week 12: number analyzed (Participants) | 19 | 12 | 16
  Week 12 | -.5 (.55) | -.2 (.44) | -.5 (.65)
  Week 16: number analyzed (Participants) | 16 | 11 | 16
  Week 16 | -.6 (.52) | -.2 (.48) | -.6 (.59)
  Week 20: number analyzed (Participants) | 16 | 15 | 15
  Week 20 | -.6 (.54) | -.5 (.69) | -.7 (.66)
  Week 24: number analyzed (Participants) | 16 | 14 | 15
  Week 24 | -.6 (.53) | -.5 (.66) | -.7 (.7)
  Week 28: number analyzed (Participants) | 15 | 14 | 14
  Week 28 | -.7 (.56) | -.5 (.63) | -.7 (.71)
  Week 32: number analyzed (Participants) | 12 | 11 | 12
  Week 32 | -.6 (.45) | -.4 (.72) | -.8 (.79)
  Week 36 | -.6 (.47) | -.2 (.59) | -.9 (.81)
  Week 40: number analyzed (Participants) | 9 | 7 | 10
  Week 40 | -.7 (.67) | -.1 (.62) | -.9 (.80)
  Week 44: number analyzed (Participants) | 7 | 5 | 7
  Week 44 | -1.0 (.62) | -.1 (.70) | -1.0 (.90)
  Week 48: number analyzed (Participants) | 6 | 6 | 7
  Week 48 | -1.1 (.61) | -.1 (.66) | -1.1 (.91)

9. Secondary Outcome: Number of Participants With Normalized Alanine Aminotransferase (ALT)
Time Frame: Baseline and at pre-specified time points up to 60 weeks
Population: Due to early termination of the study, data were not collected or analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Plasma Concentration of ABI-H0731
Time Frame: Predose on Day 1, Week 4, and Week 24 and at pre-specified time points postdose up to Week 24
Population: No ABI-H0731 PK data were collected from the ETV + Peg-IFNα group until Week 24 when they started receiving ABI-H0731.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 20 | 17 | 14
ng/mL
  Day 1, Predose: number analyzed (Participants) | 20 | 17 | 0
  Day 1, Predose | 0 (0) | 0 (0) |
  Day 1, 2 to 4 hours postdose: number analyzed (Participants) | 20 | 17 | 0
  Day 1, 2 to 4 hours postdose | 852 (552) | 1240 (550) |
  Week 2, 30 min to 2 hours postdose: number analyzed (Participants) | 20 | 16 | 0
  Week 2, 30 min to 2 hours postdose | 2130 (1190) | 1700 (802) |
  Week 4, predose: number analyzed (Participants) | 19 | 15 | 0
  Week 4, predose | 2070 (802) | 1390 (636) |
  Week 8, 30 min to 2 hours postdose: number analyzed (Participants) | 19 | 15 | 0
  Week 8, 30 min to 2 hours postdose | 2000 (780) | 1560 (559) |
  Week 12, 30 min to 2 hours postdose: number analyzed (Participants) | 19 | 12 | 0
  Week 12, 30 min to 2 hours postdose | 1920 (745) | 1650 (691) |
  Week 16, 4 to 6 hours postdose: number analyzed (Participants) | 16 | 12 | 0
  Week 16, 4 to 6 hours postdose | 2030 (610) | 2200 (855) |
  Week 20, 4 to 6 hours postdose: number analyzed (Participants) | 16 | 14 | 0
  Week 20, 4 to 6 hours postdose | 2210 (702) | 2090 (735) |
  Week 24, predose: number analyzed (Participants) | 14 | 14 | 14
  Week 24, predose | 2020 (951) | 1730 (661) | 0 (0)
  Week 24, 30 min to 2 hours postdose: number analyzed (Participants) | 14 | 14 | 14
  Week 24, 30 min to 2 hours postdose | 2070 (920) | 1580 (521) | 374 (331)

11. Secondary Outcome: Incidence of HBV Variants With Reduced Susceptibility to ABI-H0731
Time Frame: Pre-specified time points up to 60 weeks
Population: No cases met the criteria for resistance analysis.
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last study drug administration (excluding ETV), up to 60 weeks.
Description: Adverse events were regularly assessed through scheduled investigator assessment and laboratory testing.
Arm/Group | ABI-H0731 + ETV | ABI-H0731 + ETV + Peg-IFNα | ETV + Peg-IFNα
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 14/20 | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-H0731 + ETV (N=20) | ABI-H0731 + ETV + Peg-IFNα (N=17) | ETV + Peg-IFNα (N=17)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-H0731 + ETV (N=20) | ABI-H0731 + ETV + Peg-IFNα (N=17) | ETV + Peg-IFNα (N=17)
Platelet Count Decreased (Investigations) | 1 | 9 | 9
Pyrexia (General disorders) | 0 | 11 | 8
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 6 | 4
White Blood Cell Count Decreased (Investigations) | 0 | 8 | 9
Neutrophil Count Decreased (Investigations) | 1 | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 8
Aspartate Aminotransferase Increased (Investigations) | 0 | 4 | 7
Weight Decreased (Investigations) | 1 | 6 | 4
Alanine Aminotransferase Increased (Investigations) | 1 | 4 | 5
Dizziness (Nervous system disorders) | 0 | 5 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 3
Fatigue (General disorders) | 0 | 1 | 5
Headache (Nervous system disorders) | 0 | 4 | 2
Injection Site Erythema (General disorders) | 0 | 5 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 2 | 4
Blood Calcium Decreased (Investigations) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Glomerular Filtration Rate Decreased (Investigations) | 1 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 1 | 0
Amylase Increased (Investigations) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Blood Potassium Increased (Investigations) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Androgenetic Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1
Blood Cholesterol Increased (Investigations) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Blood Phosphorus Decreased (Investigations) | 1 | 0 | 0
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 0 | 1
Blood Urine Present (Investigations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 | 0 | 0
Helicobacter Infection (Infections and infestations) | 0 | 1 | 0
Hepatic Pain (Hepatobiliary disorders) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Injection Site Haemorrhage (General disorders) | 0 | 0 | 1
Injection Site Pain (General disorders) | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Mean Cell Haemoglobin Concentration Increased (Investigations) | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Pain In Extremity (General disorders) | 0 | 1 | 0
Pericoronitis (Infections and infestations) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Urinary Occult Blood Positive (Investigations) | 0 | 1 | 0
Urinary Sediment Present (Investigations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Infection (Infections and infestations) | 1 | 0 | 0
Viral Rash (Infections and infestations) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study ABI-H0731-203 was terminated early by the study Sponsor for strategic reasons to prioritize research and development efforts on finite and curative HBV therapies. As a result, not all subjects completed Week 48 and some outcome measures were impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04781647/Prot_SAP_000.pdf